CLINICAL TRIAL: NCT06567561
Title: Implementing Good Nutrition to Improve, Transform, and Enhance Firefighters' Health
Brief Title: IGNITE Firefighters' Health
Acronym: IGNITE FH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-75777; NCI-2025-01830 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Inflammation; Microbiome; Immune Function
Keywords: Cancer; Inflammation; Microbiome; Immune function
MeSH Terms: conditions — Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Food Plant-Based Diet (Experimental): Participants will be asked to consume and predominantly vegan, whole-foods diet, with the addition of fish, eggs, and fermented dairy.
  Interventions: Behavioral: Whole Foods Plant-Based Diet
- Usual Firehouse Diet (Active Comparator): Participants will be asked to consume their usual firehouse meals.
  Interventions: Behavioral: Usual Firehouse Diet

INTERVENTIONS:
Behavioral: Whole Foods Plant-Based Diet — Whole foods, predominantly plant-based diet, with the addition of fish, eggs, and fermented dairy.
  Arms: Whole Food Plant-Based Diet
Behavioral: Usual Firehouse Diet — Usual firehouse meals.
  Arms: Usual Firehouse Diet

SUMMARY:
Investigators hope to learn about potential dietary intervention strategies (specifically a whole-food, plant-based diet) that may help lower cancer markers in firefighters.

DETAILED DESCRIPTION:
The purpose of the San Francisco (SF) Firefighter's Diet Study is to determine if a diet low in processed foods, mostly plant-based, with added fermented foods, can lower the risk of cancer in firefighters. We will assess this by randomly assigning SF firefighters to either a whole-food, plant-based diet or their usual firehouse meals. Participants will be followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Active SF firefighter
* Willing to consume a plant-based diet (vegetables, fruit, whole grains, legumes, etc.)
* Willing to complete 4 clinic visits

Exclusion Criteria:

* Weight < 110 lb
* BMI >= 40
* Self-reported uncontrolled hypercholesterolemia, hypertension or diabetes
* Pregnant, lactating, or planning to become pregnant during the course of the study.
* Use of any of the following drugs/supplements within the last 2 months:

  * systemic antibiotics, antifungals, antivirals, or antiparasitics (intravenous, intramuscular, or oral);
  * corticosteroids (intravenous, intramuscular, oral, nasal or inhaled);
  * cytokines;
  * methotrexate or immunosuppressive cytotoxic agents.
* Chronic, clinically significant, or unstable (unresolved, requiring ongoing changes to medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality, as determined by medical history, Type 1 diabetes, dialysis
* History of active cancer in the past 3 years except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision
* Unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in the diet.
* Recent history of chronic excessive alcohol consumption defined as more than five 1.5-ounce servings of 80 proof distilled spirits, five 12-ounce servings of beer or five 5-ounce servings of wine per day; or > 14 drinks/week.
* Any confirmed or suspected condition/state of immunosuppression or immunodeficiency (primary or acquired) including HIV infection, multiple sclerosis, and Graves' disease.
* Surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time.
* Regular/frequent use of smoking or chewing tobacco, e-cigarettes, cigars or other nicotine-containing products
* Regular use of prescription opiate pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference in IL-6 | Baseline and 8 weeks
  Difference in the 8-week change from baseline in IL-6 between the whole-food plant-based vs. usual diet groups.

SECONDARY OUTCOMES:
Difference in Glyc a | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Glyc a between the whole-food plant-based vs. usual diet groups.
Difference in C-Reactive Protein (CRP) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in C-Reactive Protein (CRP) between the whole-food plant-based vs. usual diet groups.
Difference in Interleukin-10 (L-10) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Interleukin-10 (IL-10) between the whole-food plant-based vs. usual diet groups.
Difference in Tumor Necrosis Factor-alpha (TNF-alpha) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Tumor Necrosis Factor-alpha (TNF-alpha) between the whole-food plant-based vs. usual diet groups.
Difference in Cytokines and Inflammatory Proteins | Baseline and 8 weeks
  Difference in the 8-week change from baseline in a panel of cytokines and inflammatory proteins using the NUcleic acid Linked Immuno-Sandwich Assay (NULISA™) between the whole-food plant-based vs. usual diet groups.
Difference in Calprotectin | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Calprotectin between the whole-food plant-based vs. usual diet groups.
Difference in 8-hydroxy-2'-deoxyguanosine (8-OH-dG) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in 8-hydroxy-2'-deoxyguanosine (8-OH-dG) between the whole-food plant-based vs. usual diet groups.
Difference in Lipid Peroxidation | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Lipid Peroxidation between the whole-food plant-based vs. usual diet groups, using the Thiobarbituric acid-reactive substance (TBARS) assay.
Difference in Protein Carbonyl (protein oxidation) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Protein Carbonyl (a measure of protein oxidation) between the whole-food plant-based vs. usual diet groups, using the enzyme-linked immunosorbent assay (ELISA).
Difference in Fasting Glucose | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Fasting Glucose between the whole-food plant-based vs. usual diet groups.
Difference in Fasting Insulin | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Fasting Insulin between the whole-food plant-based vs. usual diet groups.
Difference in Low-Density-Lipoprotein Cholesterol (LDL) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Low-Density-Lipoprotein Cholesterol (LDL) between the whole-food plant-based vs. usual diet groups.
Difference in High-Density-Lipoprotein Cholesterol (HDL) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in High-Density-Lipoprotein Cholesterol (HDL) between the whole-food plant-based vs. usual diet groups.
Difference in Triglycerides (TRGs) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Triglycerides (TRGs) between the whole-food plant-based vs. usual diet groups.
Difference in Telomeres | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Telomeres between the whole-food plant-based vs. usual diet groups.
Difference in Epigenetic Age | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Epigenetic Age between the whole-food plant-based vs. usual diet groups, assessed by Epigenetic Clocks.
Difference in Gut Microbiome Composition | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Gut Microbiome Composition between the whole-food plant-based vs. usual diet groups, assessed by Metagenomic Sequencing.
Difference in Metabolomic Profiles | Baseline and 8 weeks
  Difference in the 8-week change from baseline in Gut Microbiome Composition between the whole-food plant-based vs. usual diet groups, assessed by assessed by Targeted and Untargeted Metabolomics
Difference in 4-hydroxynonenal (HNE) | Baseline and 8 weeks
  Difference in the 8-week change from baseline in 4-hydroxynonenal (HNE) between the whole-food plant-based vs. usual diet groups.
Difference in body composition | Baseline and 8 weeks
  Difference in the 8-week change from baseline in body composition between the whole-food plant-based vs. usual diet groups, as assessed by dual energy x-ray absorptiometry scan (DEXA) scans.
Difference in weight | Baseline and 8 weeks
  Difference in the 8-week change from baseline in weight between the whole-food plant-based vs. usual diet groups.
Difference in systolic blood pressure | Baseline and 8 weeks
  Difference in the 8-week change from baseline in systolic blood pressure between the whole-food plant-based vs. usual diet groups.
Difference in diastolic blood pressure | Baseline and 8 weeks
  Difference in the 8-week change from baseline in diastolic blood pressure between the whole-food plant-based vs. usual diet groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description and sign up — https://med.stanford.edu/nutrition/research/current-studies/ignite-firefighters--health.html